CLINICAL TRIAL: NCT01037686
Title: Exploring the Effect of Electrode Implantation for DBS on Brain Function During Rest and During Semantic Verbal Fluency Task Using SPECT With Tc-ECD
Brief Title: The Effect of Electrode Implantation for Deep Brain Stimulation (DBS) on Brain Function Using Single Photon Emission Computed Tomography (SPECT) With Technetium-99m-ethyl Cysteinatedimer (Tc-ECD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Sharon Hassin, principal investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-05-3972-SH-CTIL
Record Dates: First submitted 2009-09-29; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation
Keywords: PD; DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD, DBS, healthy controls (Other): Patients with idiopathic PD before or after DBS surgery (during on or off-stimulation) and healthy controls.
  Interventions: Radiation: Injection of 15mCi of Tc-ECD and scanning by SPECT camera; Behavioral: Semantic verbal fluency task performance; Device: Turning off the stimulator

INTERVENTIONS:
Radiation: Injection of 15mCi of Tc-ECD and scanning by SPECT camera — All subjects (PD patients with or without DBS and healthy controls) will be injected with 15mCi of Tc-ECD and afterwards will be scanned by an Irix SPECT camera.
Behavioral: Semantic verbal fluency task performance — All Subjects (PD patients with or without DBS and healthy controls) before one of the two scans will perform the semantic verbal fluency task during the Tc-ECD uptake for 9 minutes. Before the other scan subjects will be at rest.
Device: Turning off the stimulator — For PD patients treated with DBS, the neurologist will turn off the stimulator after the injection of Tc-ECD for ten minutes and then turn it back on.

SUMMARY:
The goal of this study is to explore the effect of subthalamic nucleus (STN)-DBS surgery and stimulation in PD (Parkinson's disease) patients on regional cerebral blood (CBF) flow during cognitive task performance or at rest.

DETAILED DESCRIPTION:
In this study subjects undergo SPECT scans for CBF mapping. PD patients before the surgery and healthy controls undergo two scans. PD patients after the surgery undergo four scans. PD patients who undergo two scans before the surgery, undergo only two scans after the surgery.

Uptake of Tc-ECD, a CBF radiotracer, is done in the following conditions:

* For PD patients before the surgery - during the performance of the semantic verbal fluency task or at rest (total of 2 scans).
* For PD patients after the surgery- during the performance of the semantic verbal fluency task or at rest, either at on-stimulation or off-stimulation condition (total of 4 scans). The stimulator is turned off by the neurologist for 10 min.
* PD patients before and after the surgery- during performance of the semantic verbal fluency task or at rest before the surgery and during performance of the semantic verbal fluency task or at rest after the surgery only at off-stimulation condition (Total of 4 scans).
* Healthy controls - during the performance of the semantic verbal fluency task or at rest (total of 2 scans).

Following the Tc-ECD injection, the subjects are scanned by Irix SPECT camera for 15min.

Scans are analyzed and the regional CBF is measured using imaging software. Statistical analysis is done to discover the effect of the surgery, stimulation and the disease on blood flow at rest and during task performance. In addition, differences between groups in number of words produced during the task are also statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Progressive idiopathic PD
* For control group - age-matched to study groups

Exclusion Criteria:

* Progressive dementia or other psychiatric disorders
* Other neurological conditions
* Other physical disease
* Intolerance of "off stimulation" state
* Involuntary head motions
* Hearing deficits

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
CBF values in different brain regions | 3 months to 2 years post-surgery

SECONDARY OUTCOMES:
Number of words produced in the semantic fluency task | 3 months to 2 years post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Clinic, Sheba Medical Center, Ramat Gan, Israel